CLINICAL TRIAL: NCT03633136
Title: Improving Health Outcomes of Kidney Recipients: A Randomized Controlled Trial of a Pre-Transplant Education Intervention
Brief Title: A Randomized Controlled Trial of a Pre-Transplant Education Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Authority - Regina Area (Other); Southern Alberta Transplant Program (Unknown); Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Principal Investigator, Holly Mansell, Associate Professor, College of Pharmacy and Nutrition, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 99302
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplant; Patient Education; Quality of Life
Keywords: video; patient education

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard education (No Intervention): Standard of care education provided at each transplant center
- electronic video education (Experimental): Standard education along with home-based video education. The videos will be initially viewed in the following order: Video 1: Introduction; Video 2: The Kidney; Video 3: Assessment and Waitlist; Video 4: Operation and Recovery; Video 5: Medications; Video 6: Your New Life. After the series has been viewed in its entirety one time, participants will be able to replay a specific video as often as desired.
  Interventions: Behavioral: electronic video education

INTERVENTIONS:
Behavioral: electronic video education — Solid Organ Transplantation: An Educational Mini-Series for Patients consists of 6 videos ranging in length between 3 and 23 minutes, and has been developed according to best practice for designing education for patients with end-stage renal disease pursuing transplant. Each video outlines a subsequent stage of the transplant process, featuring an animated character embarking on a transplant journey. Animated segments illustrate difficult concepts for patients with poor health literacy, and patient narratives keep the content relevant and culturally inclusive. The educational intervention was developed with experts in medication adherence, video education, motivational psychology, cultural education (First Nations perspective), healthcare providers, and most importantly patients.
  Other Names: Solid Organ Transplantation: An Educational Mini-Series for Patients
  Arms: electronic video education

SUMMARY:
A multi-center, randomized, controlled clinical trial will be conducted to test the effectiveness of a home-based video intervention on improving kidney transplant candidate's knowledge, self-efficacy, quality of life, beliefs in medications, and education satisfaction as compared to usual care.

DETAILED DESCRIPTION:
Kidney transplantation is the best treatment for most patients with end-stage kidney disease, but it is an extremely complicated process. To become active on the transplant waitlist, patients must learn new information, navigate the healthcare system and undergo several specialized tests. After the transplant, another set of challenges emerge. Transplant recipients must commit to lifelong therapy with immunosuppressive medications and adapt to lifestyle changes. Up to half of all patients have difficulty taking the medications as prescribed, which can lead to transplant rejection, kidney loss, and death. The transplant process is challenging and confusing; however, increasing education and support to transplant candidates demands greater use of care providers' time and resources in a health care system that is already stretched.

A patient-oriented video series has been developed according to best practices for transplant education, featuring an animated character embarking on a transplant journey. Animated segments illustrate difficult concepts for patients with poor health literacy, and patient narratives provide support and encouragement.

A multi-center, randomized, controlled clinical trial will be conducted to test the effectiveness of a home-based video intervention on improving kidney transplant candidate's knowledge, self-efficacy, quality of life and beliefs in medications as compared to usual care. Participants will be randomized (1:1) to the control group, or the intervention group, who will be provided access to the video series, in addition, to standard of care. Differences in changes in transplant knowledge, self-efficacy, beliefs about medicines, quality of life, and education satisfaction will be evaluated by a pre-and post-intervention survey. A thorough assessment of video-viewing habits and satisfaction with the intervention will provide insight on the feasibility of expanding home-based education to other health settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* can speak and understand and read English
* are being assessed or wait-listed for kidney transplantation

Exclusion Criteria:

* do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Change in transplant knowledge score between the intervention and control groups as measured by the Kidney Transplant Understanding Tool (K-TUT) | 1 month
  Measured by the Kidney Transplant Understanding Tool (K-TUT) (self-reported electronic survey). The K-TUT consists of 9 true/false and 13 multiple-choice questions, and scores are based on the number correct answers [YES/ NO format] of 69 items.

SECONDARY OUTCOMES:
Difference in self-efficacy between the intervention and control group as measured by the Generalized Self Efficacy Scale (GSE) | 1 month
  Measured by the Generalized Self Efficacy Scale (GSE) (self-reported electronic survey).The GSE measures an individual's self-beliefs in their ability to cope with various demands in life. It is a 10-item psychometric scale with a score for each item ranging from 1 to 4. The scores are summed and a higher score indicates stronger patient beliefs in self-efficacy.
Difference in quality of life between the intervention and control group as measured by the Short Form-12 (SF-12) | 1 month
  Measured by the Short Form-12 (SF-12) (self-reported electronic survey). The SF-12 is a 12-item psychometric scale that measures functional health and well-being. Responses are indicated on a likert scale and aggregated into two sub scales; the mental component summary (MCS) and the physical component summary (PCS). The scores are converted to adjusted norm-based values of a healthy individual with a midpoint score of 50 indicating average health comparable to norm values.
Difference in beliefs of medicine between the intervention and control group as measured by the Beliefs of Medicine Questionnaire (BMQ) | 1 month
  Measured by the Beliefs of Medicine Questionnaire (BMQ) (self-reported electronic survey). The BMQ is an 18-item psychometric questionnaire which consists of two subscales. The BMQ-Specific assesses perceptions of medication prescribed for personal use, while the BMQ-General assesses beliefs about medications in general. The BMQ-General can be further classified into domain of General-Harm and General-Overuse. Items are scored on a 5-point likert scale, with higher score indicating stronger beliefs in each subscale.
Difference in education satisfaction between the intervention and control group as measured by self-reported electronic survey | 1 month
  Measured by self-reported electronic survey

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Southern Alberta Transplant Program, Calgary, Alberta
  - Saskatchewan Transplant Program, Regina, Saskatchewan
  - Saskatchewan Transplant Program, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: project website — https://words.usask.ca/transplant/
- See also: Study Results — https://journals.lww.com/transplantationdirect/fulltext/2021/10000/a_randomized_controlled_trial_of_a_pretransplant.8.aspx